CLINICAL TRIAL: NCT07170280
Title: Radiological and Functional Evaluation of Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures: A Prospective Cohort Study
Brief Title: Evaluation of Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures
Acronym: Infrapectineal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahmoud Fahmy (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Fahmy, associate professor of orthopaedic surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-350-2021
Record Dates: First submitted 2025-08-29; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Trauma (Including Fractures)
Keywords: Acetabular fracture; Surgical fixation; Quadrilateral plate; Ilioinguinal approach
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Quadrilateral plate acetabular fractures are complex injuries that present challenges in achieving stable fixation due to their anatomical location and high risk of medial displacement. The direct infrapectineal plate, applied via the ilioinguinal approach, offers a biomechanically stable construct for buttressing the medial acetabular wall.
  This prospective cohort study enrolled 25 patients aged 18-64 years with acute quadrilateral plate acetabular fractures between January 2021 and January 2024. Patients with pathological fractures, pre-existing ipsilateral hip disease, or delayed presentation (>4 weeks) were excluded.
  The surgical procedure involved direct infrapectineal plating through the ilioinguinal approach. Radiological outcomes were measured using the Matta scoring system, and functional results were assessed with the Merle d'Aubigné and Postel scoring system at a mean follow-up of 14.7 months. Secondary measures included operative time, blood loss, hospital stay, and compl
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiological and Functional Evaluation of Direct Infrapectineal Plating in Quadrilateral Plate Aceta (Other): Quadrilateral plate acetabular fractures are complex injuries that present challenges in achieving stable fixation due to their anatomical location and high risk of medial displacement. The direct infrapectineal plate, applied via the ilioinguinal approach, offers a biomechanically stable construct for buttressing the medial acetabular wall.
  This prospective cohort study enrolled 25 patients aged 18-64 years with acute quadrilateral plate acetabular fractures between January 2021 and January 2024. Patients with pathological fractures, pre-existing ipsilateral hip disease, or delayed presentation (>4 weeks) were excluded.
  The surgical procedure involved direct infrapectineal plating through the ilioinguinal approach. Radiological outcomes were measured using the Matta scoring system, and functional results were assessed with the Merle d'Aubigné and Postel scoring system at a mean follow-up of 14.7 months. Secondary measures included operative time, blood loss, hospital stay, and comp
  Interventions: Procedure: Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures: A Prospective Cohort Study

INTERVENTIONS:
Procedure: Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures: A Prospective Cohort Study — This study aims to evaluate the outcomes of direct infrapectineal plate fixation in patients with quadrilateral plate acetabular fractures. A total of 25 adult patients with acute fractures were enrolled between 2021 and 2024 at a university-affiliated hospital. All patients underwent surgical fixation through the ilioinguinal approach. Radiological results were assessed using the Matta scoring system, and functional outcomes were evaluated using the Merle d'Aubigné and Postel scoring system. The study further assessed complication rates, operative time, intraoperative blood loss, and hospital stay.

SUMMARY:
This study aims to evaluate the outcomes of direct infrapectineal plate fixation in patients with quadrilateral plate acetabular fractures. A total of 25 adult patients with acute fractures were enrolled between 2021 and 2024 at a university-affiliated hospital. All patients underwent surgical fixation through the ilioinguinal approach. Radiological results were assessed using the Matta scoring system, and functional outcomes were evaluated using the Merle d'Aubigné and Postel scoring system. The study further assessed complication rates, operative time, intraoperative blood loss, and hospital stay.

DETAILED DESCRIPTION:
Quadrilateral plate acetabular fractures are complex injuries that present challenges in achieving stable fixation due to their anatomical location and high risk of medial displacement. The direct infrapectineal plate, applied via the ilioinguinal approach, offers a biomechanically stable construct for buttressing the medial acetabular wall.

This prospective cohort study enrolled 25 patients aged 18-64 years with acute quadrilateral plate acetabular fractures between January 2021 and January 2024. Patients with pathological fractures, pre-existing ipsilateral hip disease, or delayed presentation (>4 weeks) were excluded.

The surgical procedure involved direct infrapectineal plating through the ilioinguinal approach. Radiological outcomes were measured using the Matta scoring system, and functional results were assessed with the Merle d'Aubigné and Postel scoring system at a mean follow-up of 14.7 months. Secondary measures included operative time, blood loss, hospital stay, and complication profile.

Preliminary results showed that anatomical reduction was achieved in 64% of patients, with excellent or good functional results in 68%. The complication rate was low, with only one case of deep infection requiring implant removal.

The study concludes that infrapectineal plating provides stable fixation with favorable functional and radiological outcomes for quadrilateral plate acetabular fractures.

ELIGIBILITY:
Inclusion Criteria:Adults aged 18-64 years.

Acute quadrilateral plate acetabular fractures (≤3 weeks from injury).

Medically fit for surgery under general or regional anesthesia.

Patients willing to participate and provide informed consent. -

Exclusion Criteria:Pathological fractures (e.g., metastatic or metabolic).

Pre-existing ipsilateral hip pathology affecting radiological or functional outcomes.

Delayed presentation: injury >4 weeks before surgery.

Medical contraindications to surgery (e.g., unstable comorbidities).

Polytrauma patients with hemodynamic instability.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Radiological and Functional Evaluation of Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures: A Prospective Cohort Study | 4 years
  Primary Outcome Measures
  Description: Radiographic assessment using the Matta scoring system at long-term follow-up.
  Time Frame: monthly till 4 years postoperatively
  Description: Postoperative anteroposterior and Judet pelvic radiographs assessed using the Matta scoring system. Reduction quality classified as anatomical (0-1 mm displacement), imperfect (2-3 mm), or poor (>3 mm).Radiological outcome at long-term follow-up
  Unit of Measure: Number of patients per reduction category

SECONDARY OUTCOMES:
Radiological and Functional Evaluation of Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures: A Prospective Cohort Study | 4 years
  Functional outcome (Merle d'Aubigné and Postel scoring system)
  Time Frame: monthly till 4 years postoperatively Description: Functional evaluation of hip pain, mobility, and walking ability using the Merle d'Aubigné and Postel scoring system. Outcomes categorized as excellent, good, fair, or poor.
  Unit of Measure: Number of patients per functional category

OTHER OUTCOMES:
Radiological and Functional Evaluation of Direct Infrapectineal Plating in Quadrilateral Plate Acetabular Fractures: A Prospective Cohort Study Primary Outcome Measures | 4 years
  Complication rate
  Time Frame: Within 4 years postoperatively
  Description: Incidence of postoperative complications including infection, thromboembolic events, implant-related issues, or loss of fixation.
  Unit of Measure: Number of patients with complications

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (e.g., baseline demographics, intraoperative details, postoperative outcomes, functional and radiological scores) that underlie the results reported in the publication will be shared. No direct identifiers will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting materials will be available beginning 12 months after publication of the primary results and will remain available for 36 months thereafter.
Access Criteria: Data will be available to qualified researchers with methodologically sound proposals. Requests should be submitted to the corresponding author. Access will be granted following review and approval of the request and execution of a data use agreement. Data will be provided in a secure format (e.g., password-protected files).
URL: https://medicine.cu.edu.eg